CLINICAL TRIAL: NCT05509465
Title: Usability and Acceptability of an Ergonomic Chinrest With or Without Shoulder Rest During Violin Playing: a Feasibility Study
Brief Title: Using an Ergonomic Chinrest With or Without Shoulder Rest During Violin Playing: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Axel Muusfeldts fond (Unknown); Region of Southern Denmark (Other); Sygekassernes Helsefond (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 10.990
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Ergonomics
Keywords: Feasibility; Violin playing; ergonomic chinrest; performance

STUDY DESIGN:
Intervention Model Description: The two intervention groups (EC+ and EC-) consist of the same participants. Every day the same participants have to divide their violin playing time equally between playing with EC+ and EC-. Each day the order of the interventions is decided by the participants.
Masking Description: This study is open label, meaning that no masking occurs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ergonomic chinrest used with low shoulder rest (EC+) (Experimental): Participants will play the violin using the ergonomic chinrest with a low Kun Super shoulder rest (EC+) for a two-week period to test its usability and acceptability. Each day participants have to use half of their playing time with EC+.
  Interventions: Device: Ergonomic chinrest used with a low Super Kun shoulder rest
- Ergonomic chinrest used without shoulder rest (EC-) (Experimental): Participants will play the violin using the ergonomic chinrest without a shoulder rest for a two-week period to test its usability and acceptability. Each day participants have to use half of their playing time with EC-.
  Interventions: Device: Ergonomic chinrest

INTERVENTIONS:
Device: Ergonomic chinrest — The novel ergonomic chinrest (Kréddle®, Wyoming, US) is fully adjustable to accommodate each violinist's body type and performance style: regarding height, rotation and tilting.
  Arms: Ergonomic chinrest used without shoulder rest (EC-)
Device: Ergonomic chinrest used with a low Super Kun shoulder rest — The novel ergonomic chinrest (Kréddle®, Wyoming, US) is fully adjustable to accommodate each violinist's body type and performance style: regarding height, rotation and tilting. The low Super Kun shoulder rest has been adjusted to be in the lowest position for all legs attached to the violin before the violinists received it. All participants was told not to adjust the shoulder rest but adjust the chinrest.
  Arms: Ergonomic chinrest used with low shoulder rest (EC+)

SUMMARY:
A one-arm feasibility study was conducted to test if violinists would accept to play with an identified ergonomic chinrest (EC) with the brand name Kréddle every day for two weeks. Every day the participants had to divide their total playing time equally between EC+ (ergonomic chinrest with shoulder rest) and EC- (ergonomic chinrest without shoulder rest) each day.

DETAILED DESCRIPTION:
This study is testing the feasibility (usability and acceptability) of a two-week familiarization period where violinists usually playing with a shoulder rest had to play their violin with an ergonomic chinrest (EC) with (EC+) and without a shoulder rest (EC-).

Primary outcomes were compliance, adherence, usability and acceptability of the familiarization period.

Prior the familiarization period each violinist received the chinrest (Kréddle) and a shoulder rest (Kun Super rest violin 4/4) and had to follow instructions given through three introduction videos.

The included violinists received a web questionnaire (QA) before and after the familiarization period. This period is unsupervised with the EC (ergonomic chinrest). Every day each violinist should equally divide their total playing time between playing without shoulder rest (EC-) and the other half with the shoulder rest (EC+) with the EC. A diary was answered each day containing different questions in regard to playing hours and usability.

The reporting in this study adheres to the CONSORT 2010 extension for pilot and feasibility trials.

When this study was initiated, we aimed at a sample size of 10-12 as a rule of thumb for a pilot/feasibility study. However, due to the corona pandemic and the many national restrictions including keeping distance, seeing only a few people, getting tested for the virus and staying at home, if possible, this number could not be reached. Even though the study was planned to include more participants the result from this small study is pointing in one direction, which is supported in a previous study as well.

ELIGIBILITY:
Inclusion Criteria:

* Writing and speaking Danish or English fluently. Participants had to be trained violinists who could play the protocol classical repertoire and without a permanent employment contract in a Danish symphony orchestra.

Exclusion Criteria:

* Trauma on the upper cervical spine or upper extremities within the previous year, previous or planned shoulder/neck operation, life-threatening health disorders, pacemaker or severe eczema on neck and upper extremities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Usability | Two weeks
  Self-reported information about the usability of the EC- and EC+ was obtained by asking questions about perceived performance, comfort, and sound experience, as well as adjustment and confidence level. Furthermore, if the instructions videos given prior to the familiarization period were usable.
Acceptability | Two weeks
  Every day each violinist was encouraged to write feedback in the diary about using EC+, EC- and about the intervention. The descriptions and comments were categorized into comments about using EC-, EC+ or general comments; the response was grouped as positive or negative feedback.
Adherence | Two weeks
  Adherence to the protocol was recorded from the self-administrated two-week diary. The violinist had to answer a small questionnaire and play each day with one of the settings. Adherence is counted as numbers of days played with the different settings out of the two weeks given.
Compliance | Two weeks
  Compliance for playing with EC- and EC+ was reached if the violinist managed to play minimum 25% out of total playing time with each of both settings. If compliance was <25% it was considered that it would be a problem to use the setting

SECONDARY OUTCOMES:
Neck movement was recorded by the device called ViMove. | Two weeks
  Neck movement data was collected with ViMove measured in degrees of movement in three anatomical planes. This was done after the two weeks and the violinists had to play with both EC and their own preferred chinrest (usual). These data were collected to make a sample size estimation for a planned larger study.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Søgaard, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No